CLINICAL TRIAL: NCT05466591
Title: Acute Rule Out of Non ST-segment Elevation Acute Coronary Syndrome in the (Pre)Hospital Setting by HEART Score Assessment and a Single Point-of-care Troponin
Brief Title: Pre-hospital Rule-out of Acute Coronary Syndrome
Acronym: ARTICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Cyril Camaro, Principal Investigator, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NL 66755.091.18; NTR7346 (Registry Identifier: Netherlands Trial Register); NTR7346 (Registry Identifier: International Clinical Trials Registry Platform); 852001942 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Point-of-care troponin; HEART score; Acute Coronary Syndrome; Myocardial infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: The patients are randomised to 1) pre-hospital rule-out with POC troponin measurement (intervention group) and 2) direct transfer to the ED (standard care group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The clinical events are blindly adjudicated by an independent Clinical Events Committee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-hospital rule-out strategy (Experimental): Patients undergo a point-of-care troponin T measurement. If troponin is low, an acute coronary syndrome is considered ruled-out and the care for the patient is transferred to the general practitioner. If troponin is elevated, the patient is immediately transported to the emergency department.
  Interventions: Diagnostic Test: Pre-hospital rule-out strategy
- Emergency department rule-out strategy (No Intervention): According to standard care, the patients are immediately transported to the emergency department.

INTERVENTIONS:
Diagnostic Test: Pre-hospital rule-out strategy — Point-of-care troponin measurement for pre-hospital rule-out of acute coronary syndrome
  Arms: Pre-hospital rule-out strategy

SUMMARY:
Patients with chest pain suspected for non ST-segment elevation acute coronary syndrome (NSTE-ACS) are routinely transferred to the emergency department (ED). A point-of-care (POC) troponin measurement might enable ambulance paramedics to identify low-risk patients in whom ED evaluation is not necessary. The ARTICA trial aims to assess the healthcare cost reduction and safety of a pre-hospital rule-out strategy using a single POC troponin measurement.

DETAILED DESCRIPTION:
Patients with chest pain suspected of a NSTE-ACS are screened by ambulance paramedics. The HEAR score (HEART score without the Troponin component) is assessed and patients with a HEAR score of ≤3 are included. The patients are randomised to 1) pre-hospital rule-out with POC troponin measurement (intervention group) and 2) direct transfer to the ED (standard care group). Primary outcome is healthcare costs after 30 days.

ELIGIBILITY:
Inclusion criteria:

* Age at least 18 years; male ánd female
* All out-of-hospital patients with chest pain or symptoms suggestive of ACS initially visited by an ambulance with an indication for transfer to a hospital to evaluate and rule out ACS
* Symptom duration for at least two hours
* Modified HEAR(T) score less or equal than 3
* A point of care troponin below the upper reference limit (for patients stratified to pre-hospital management by the general practitioner)
* The patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion criteria:

* Electrocardiographic ST-segment elevation
* Patients presenting an obvious non-cardiac cause for the chest complaints who need evaluation at an emergency department, e.g. trauma, pneumothorax, sepsis, etc.
* Patients in comatose state, defined as an Glascgow coma scale (GCS) <8
* Patients with known cognitive impairment
* Pregnancy or intention to become pregnant during the course of the study
* Patients presenting cardiogenic shock, defined as: systolic blood pressure <90 mmHg and heart rate >100 beats per minute and peripheral oxygen saturation <90% (without oxygen administration)
* Patients presenting with syncope
* Patients presenting with signs of heart failure
* Patients presenting with heart rhythm disorders and second or third degree atrioventricular block
* Patients with known end-stage renal disease (dialysis and/or glomular filtration rate (GFR) < 30 ml/min)
* Patients without a pre-hospital 12-lead ECG performed or available
* Patients suspicious of aortic dissection or pulmonary embolism
* Patients with confirmed acute myocardial infarction, percutaneous coronary intervention or coronary artery bypass grafting <30 days prior to inclusion
* Communication issues with patient/language barrier
* Decision of a present general practitioner to evaluate the patient at the emergency department (ED)
* Decision of the consultant cardiologist to evaluate patient at the ER irrespective of HEART score
* Any significant medical or mental condition, which in the Investigators opinion may interfere with the patients optimal participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 866 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2023-05-04 (Estimated)

PRIMARY OUTCOMES:
Costs from a healthcare perspective (all costs related to healthcare consumption in-hospital, all outpatient visits including diagnostic tests and general practitioner consultations) | 30 days
  Healthcare costs consist of all costs related to healthcare consumption

SECONDARY OUTCOMES:
Safety: all cause death, acute coronary syndrome, unplanned revascularisation | 30 days
  Major adverse cardiac events (all cause death, ACS, unplanned revascularisation)
Costs from a societal perspective (all health effects and changes in resource use caused by an intervention) | 30 days
  Costs from a societal perspective are defined as the sum of the healthcare costs and the costs from productivity losses.
Safety (all cause death, acute coronary syndrome, unplanned revascularisation) | 6 months
  Major adverse cardiac events (all cause death, ACS, unplanned revascularisation)
Safety (all cause death, acute coronary syndrome, unplanned revascularisation) | 12 months
  Major adverse cardiac events (all cause death, ACS, unplanned revascularisation)

CONTACTS AND LOCATIONS:
Overall Officials: Niels van Royen, MD PhD Prof, Study Chair — Radboud University Medical Center
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to researchers who were granted permission to the data by the principal investigator
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year after completion
Access Criteria: After permission

REFERENCES:
- [Derived] Aarts GWA, Camaro C, Rodwell L, Adang EMM, van Hout R, Brok G, Hoare A, de Pooter FPC, de Wit W, Cramer GE, van Kimmenade RRJ, Ouwendijk E, Rutten M, Zegers E, van Geuns RM, Gomes MER, Damman P, van Royen N. Differences in risk and costs between prehospital identified low-risk men and women with chest pain. Open Heart. 2023 Nov 27;10(2):e002390. doi: 10.1136/openhrt-2023-002390. PMID 38011992
- [Derived] Camaro C, Aarts GWA, Adang EMM, van Hout R, Brok G, Hoare A, Rodwell L, de Pooter F, de Wit W, Cramer GE, van Kimmenade RRJ, Damman P, Ouwendijk E, Rutten M, Zegers E, van Geuns RM, Gomes MER, van Royen N. Rule-out of non-ST-segment elevation acute coronary syndrome by a single, pre-hospital troponin measurement: a randomized trial. Eur Heart J. 2023 May 14;44(19):1705-1714. doi: 10.1093/eurheartj/ehad056. PMID 36755110
- See also: Study website — http://articatrial.nl/en/artica-2/